CLINICAL TRIAL: NCT03158116
Title: A-PACT: The Use of Inhaled Aztreonam to Eliminate or Decrease the Bacterial Burden of Pseudomonas Aeruginosa in Children With a Tracheostomy Tube.
Brief Title: The Use of Inhaled Aztreonam in Children With a Tracheostomy Tube and Pseudomonas
Acronym: A-PACT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB application expired.
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 2016-009
Record Dates: First submitted 2017-04-18; First posted 2017-05-17 (Actual); Results first posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Tracheostomy Infection
Keywords: tracheostomy tube; Pseudomonas aeruginosa
MeSH Terms: conditions — Pseudomonas Infections

STUDY DESIGN:
Intervention Model Description: two-center, prospective, case control clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (Experimental): All participants will be receiving the study drug
  Interventions: Drug: Inhaled Aztreonam

INTERVENTIONS:
Drug: Inhaled Aztreonam — Inhaled antibiotic with anti-pseudomonal properties

SUMMARY:
This is a prospective, case-control clinical trial using inhaled Aztreonam (AZLI) in pediatric patients with a tracheostomy tube colonized with Pseudomonas aeruginosa. The aim of the study is to see if AZLI being taken in a one month on / one month off cycle over the course of a year can decrease the need for systemic antibiotics and/or hospitalizations.

DETAILED DESCRIPTION:
Inhalation aztreonam (AZLI) is an aerosolized formulation of the monobactam antibiotic aztreonam with lysine as a synthetic substance in place of arginine. This substitution was made as arginine, which is in the intravenous (IV) formulation of aztreonam, can cause airway inflammation as seen in patients with cystic fibrosis when aerosolized. There have been several published studies on the efficacy and adverse effects of aerosolized aztreonam in CF patients. Two placebo-controlled studies of AZLI revealed a benefit in patients with CF and colonization with PsA. AIR-CF1 revealed that a 28-day course of AZLI given three times daily (TID) resulted in improved respiratory symptoms. They measured this improvement by using a cystic fibrosis questionnaire (CFQ-R), measuring forced expiratory volume in 1 second (FEV 1), and measuring bacterial density in sputum. AIR-CF2 demonstrated that a 28-day course of AZLI followed by a 28-day course of Tobramycin Inhaled Solution (TIS) delayed the time to the need for additional inhaled or systemic anti-pseudomonal antibiotics. They also used the CFQ-R and measured FEV1 and found improvement in both when compared to placebo. In AIR-CF3, an open-label 18-month study was conducted to evaluate the efficacy of AZLI using a month on/month off cycle, and to observe long-term effects of the drug. This protocol found that AZLI did have a long-term suppressive effect on PsA as there was a persistent reduction in Pseudomonas CFUs from baseline each month of the study. As expected, the decreases in bacterial density were consistently occurring during on months; and during off months, the density increased toward baseline. Thrice-daily dosing appeared more efficacious than twice-daily dosing. This was attributed to the mode of action of aztreonam, as bacterial killing is dependent on time above the MIC (minimal inhibitory concentration). Adverse events include: cough, respiratory tract congestion, pharyngolaryngeal pain, nasal congestion, dyspnea, hemoptysis, rhinorrhea, wheezing, chest discomfort, crackles lung, pulmonary function testing decreased, non-cardiac chest pain, sinus congestion, sinus headache, dyspnea exacerbated, exertional dyspnea.

Antibiotics currently on the market as inhaled antibiotics include tobramycin (TOBI), polymyxin E (Colistin), and aztreonam (Cayston). Studies of all of these have shown clinical benefits in those with Cystic Fibrosis. Given these findings, there is a growing interest in the use of inhaled antibiotics in other disease processes in which subjects become colonized with bacteria in the lower respiratory tract.

The investigators propose a two-center, prospective, case control clinical trial on the use of inhaled aztreonam (AZLI) in pediatric patients ages 7-21 years with a tracheostomy who have had one of their previous 3 tracheostomy aspirate cultures positive for PsA. Their past history in the previous year of requirement for systemic antibiotics will be used for each subject as the historical control. A tracheostomy aspirate culture will be collected upon initiation of the study. The investigators will subsequently start the participants on AZLI on a one month on/one month off schedule. Tracheal aspirate cultures will continue to be collected quarterly (every 3 months), and the bacterial density will be used for analysis. Goal is to see if there is a decrease need for systemic antibiotics for PsA infection.

ELIGIBILITY:
Inclusion Criteria:

* o Age: 7 - 21 years old

  * Currently has a tracheostomy tube
  * One of previous 3 tracheostomy tube aspirate cultures positive for Pseudomonas aeruginosa
  * Non-smoker
  * Ability of parent to provide informed consent, as evidenced by signing a copy of the consent form approved by the Institutional Review Board of the subject's respective study institution.
  * Written assent for children 7-17 years of age.
  * Informed consent for children ages 18-21, as evidence by signing a copy of the consent form approved by the Institutional Review Board of the subject's respective study institution.

Exclusion Criteria:

* o History of immunodeficiency

  * History of cystic fibrosis. Primary ciliary dyskinesia, or bronchiectasis
  * History of tuberculosis
  * History of positive culture for Burkholderia cepacia
  * Use of inhaled antibiotics in the last 6 months

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachna Wadia, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 11.6 [8 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 1
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 1
  Race: White | 0
  Race: More than one race | 0
  Race: Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decreased Need for Systemic Antibiotics While on the Study Drug
Description: Number of participants with a reduced number of days of systemic antibiotics needed after participant starts using the study drug. (compare 1 year prior to starting study drug to the 1 year while patient is on the study drug)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

2. Secondary Outcome: Bacterial Density
Description: See if bacterial density of Pseudomonas is decreased or eliminated with the study drug (will compare all cultures from the year prior to starting the trial to the year during the trial)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Tracheostomy Tube Type
Description: to see if there is a difference in how effective the study drug is depending on what type of trach tube the subject has. Will assess this by looking at the Pseudomonas bacterial density from the tracheostomy tube cultures from the year prior to starting the study drug and compare to the year while on the study drug.
Time Frame: 1 year
Population: Because all participants had the Bivonia trach tube, this outcome measure could not be evaluated.
Arm/Group | Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With a Decreased Number of Hospital Admissions
Description: Number of participants with a reduced number of hospital admissions the year prior to starting the study drug compared to the year while taking the study drug.
  Can study drug decrease number of hospital admissions form the year prior to starting the study drug compared to the year while taking the study drug?
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Number of Participants With a Decrease in the Duration of Hospitalizations
Description: Can the study drug decrease the duration of hospitalizations from the year prior to starting the study drug compared to the year while taking the study drug?
Time Frame: 1 year
Population: None of the subjects required hospitalization for a primary respiratory illness during the study visit, so hospital stay duration could not be compared.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The study has limitations with the primary one being it is a very small study. The intention was to have a larger study multi-center study. However, due to multi-site institutional research logistics and administrative bureaucracy, expanding the study was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT03158116/Prot_SAP_000.pdf